CLINICAL TRIAL: NCT05607173
Title: A Multicentric, Open-label, Non-randomized, Pharmacokinetic and Tolerability Study of Fexinidazole Given as an Oral Single 1200 mg Dose in Participants With Mild and Moderate Hepatic Impairment, and in Matched Participants With Normal Hepatic Function
Brief Title: A Pharmacokinetic and Tolerability Study of Fexinidazole in a Single Oral Dose in Adult Participants With Mild and Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: POP17145; U1111-1266-5794 (Registry Identifier: ICTRP); 2021-004580-27 (EudraCT Number)
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Function Abnormal
MeSH Terms: conditions — Liver Diseases | interventions — fexinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Participants with mild HI (Experimental): Mild HI is defined as a total score ranging from 5 to 6, inclusive (Child-Pugh score A)
  Interventions: Drug: Fexinidazole (HOE239)
- Participants with moderate HI (Experimental): Moderate HI is defined as a total score ranging from 7 to 9, inclusive (Child-Pugh score B)
  Interventions: Drug: Fexinidazole (HOE239)
- Participants with normal hepatic function (Experimental): Participants with normal hepatic function matched to participants
  Interventions: Drug: Fexinidazole (HOE239)

INTERVENTIONS:
Drug: Fexinidazole (HOE239) — Route of administration: oral; pharmaceutical form: tablet
  Other Names: Fexinidazole Winthrop®

SUMMARY:
In human, metabolic hepatic clearance represents a significant part of the total clearance of fexinidazole and could be decreased in patients with liver impairment, leading to some overexposure, and conversely, the formation of the 2 active metabolites could be decreased, leading to decreased exposure in hepatic impairment (HI).

As there is no experience of use in patients with hepatic impairment, in fexinidazole summary of product characteristics (SmPC) approved by the European Medicines Agency (EMA), fexinidazole is contra-indicated in patients with clinical signs of cirrhosis or jaundice, and in the proposed USA product information, fexinidazole is contra-indicated in patients with liver impairment.

Therefore, FDA requested a study with the objective to evaluate the effect of mild and moderate hepatic impairment (HI) on the pharmacokinetics (PK) of fexinidazole and its 2 metabolites, as a post-marketing requirement.

DETAILED DESCRIPTION:
The duration of the study for 1 participant will be of 38 days maximum, including:

* A screening period from Day (D)-28 to D-2
* Baseline assessments on D-1
* Single dose administration on D1 and institutionalization for 6 days
* End of study (EOS): D10, or to be organized as soon as possible in case of early withdrawal

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, between 18 and 75 years of age, inclusive
* 12-lead ECG without clinically significant abnormality, in the judgment of the Investigator; normal QT interval confirmed
* Contraception (with double contraception methods) for male and female (unless postmenopausal) participants; not pregnant or breastfeeding for female participants; no sperm donation for male participants.
* Having given written informed consent prior to any procedure related to the study
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research
* Not under any administrative or legal supervision

Participants with HI

* Body weight between 50.0 and 125.0 kg, inclusive if male, and between 40.0 and 110.0 kg, inclusive if female, body mass index (BMI) between 18.00 and 34.99 kg/m2, inclusive
* Stable chronic liver disease assessed by medical history, physical examination, laboratory values
* Vital signs after 10 minutes resting in supine position within the following range [or if out of range, considered not clinically significant (NCS) by the Investigator]:

  * 95 mmHg < systolic blood pressure (SBP) < 180 mmHg
  * 45 mmHg < diastolic blood pressure (DBP) < 100 mmHg
  * 40 bpm < HR < 100 bpm
* Laboratory parameters within the acceptable range for participants with HI; however, serum creatinine should be strictly below the upper laboratory normal
* For moderate HI cohort: Child-Pugh total score ranging from 7 to 9, inclusive
* For mild HI cohort: Child-Pugh total score ranging from 5 to 6, inclusive

Matched participants with normal hepatic function

* Body weight within 15% of the mean body weight of the participants with HI to be matched, and BMI between 18.00 and 34.99 kg/m2, inclusive
* Certified as healthy by a comprehensive clinical assessment
* Vital signs after 10 minutes resting in the supine position within the following range:

  * 95 mmHg < SBP < 160 mmHg
  * 45 mmHg < DBP < 90 mmHg
  * 40 bpm < HR < 100 bpm
* Laboratory parameters within the normal range, excluding specific exceptions allowed per protocol.

Exclusion Criteria:

* Participant has clinical signs and symptoms consistent with COVID-19, e.g., fever, dry cough, dyspnea, loss of taste and smell, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening. Participant who had severe course of COVID-19
* Positive test for SARS-CoV-2
* Blood donation within 2 months before inclusion
* Postural hypotension - symptomatic or asymptomatic (decrease in SBP ≥ 30 mmHg within 3 minutes).
* Excessive consumption of beverages with xanthine bases
* COVID-19 vaccination: last administration of a vaccine within 1 week (symptom free) to 2 weeks before inclusion
* Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development
* Any participant in the exclusion period of a previous study according to applicable regulations
* Any participant who cannot be contacted in case of emergency
* Positive alcohol breath test
* Any consumption of citrus fruits or their juices within 5 days before inclusion
* Unable or not agreeing to self-complete the hospital anxiety and depression scale (HADS)
* Hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
* Positive result on anti-human immunodeficiency virus 1 and/or 2 antibodies
* Cockayne Syndrome

Participants with HI

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecological (if female), or infectious disease, or signs of acute illness
* Hepatocarcinoma
* Acute hepatitis
* Hepatic encephalopathy grade 2, 3, and 4
* Presence or history of drug hypersensitivity, or allergic disease, including active seasonal rhinitis, diagnosed and treated by a physician
* History or presence of regular use of recreational drugs or alcohol abuse within 2 years before inclusion
* Smoking more than 15 cigarettes or equivalent per day, unable to refrain from smoking over 5 cigarettes per day from D-1 and throughout the entire institutionalization
* Any significant change in chronic treatment medication within 14 days before inclusion
* Consumption of CYP450 potent inducers or inhibitors that could impact the pharmacokinetics of the investigational product
* Positive results on urine drug screen outside documented medical prescription
* Pre-existing cardiac disease, long QT syndrome, or use of drugs known to block potassium channels, prolong the QT interval and/or induce bradycardia

Matched participants with normal hepatic function

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecological (if female), or infectious disease, or signs of acute illness
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician, except seasonal rhinitis
* History or presence of regular use of recreational drugs or alcohol abuse
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking from D-1 and throughout the entire institutionalization
* Any medication (including CYP450 inducers or inhibitors, or omeprazole) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic (PD) half-life of the medication (except HRT and contraception when applicable), any vaccination within the last 28 days (except COVID-19 vaccination) and any biologics (antibody or its derivatives) given within 4 months before inclusion
* Positive result on any of the following tests: hepatitis B surface antigen, antihepatitis B core antibodies, anti-hepatitis C virus antibodies
* Positive result on urine drug screen

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Cmax for fexinidazole and metabolites M1, M2 | Day 1 to Day 6
  Maximum plasma concentration observed (Cmax)
AUC for fexinidazole and metabolites M1, M2 | Day 1 to Day 6
  Area under the plasma concentration versus time curve extrapolated to infinity (AUC)

SECONDARY OUTCOMES:
tmax for fexinidazole and metabolites M1, M2 | Day 1 to Day 6
  Time to reach Cmax (tmax)
Fexinidazole unbound fraction | Day 1 and Day 2
Fexinidazole unbound Cmaxu | Day 1 and Day 6
  Unbound maximum plasma concentration observed (Cmaxu)
Fexinidazole unbound AUCu | Day 1 and Day 6
  Unbound area under the plasma concentration versus time curve extrapolated to infinity
Number of subjects with Adverse Events (AEs) | Day 1 to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Investigational Site Number: 100-0001, Sofia, Bulgaria
- Investigational site 250-0001, Rennes, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: POP17145 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25335&tenant=MT_SNY_9011